CLINICAL TRIAL: NCT01350661
Title: Assessment of Correlation Between Five Asthma Control Questionnaires
Brief Title: Correlation Between Five Asthma Control Questionnaires
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Dr. Inge Muylle, Dr. Inge Muylle, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: B07620109010
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
Keywords: Asthma; Questionnaires
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma control level assessment

SUMMARY:
This observational study aims to assess the correlation between many questionnaires designed to assess the level of control of asthma. The five questionnaires will be submitted, at the same time and in a random order, to asthma patients. Some other parameters will be recorded (e.g. lung function, epidemiological data). The hypothesis is that the results of the questionnaires will be the same. If not, we will try to understand why.

The investigators will include 100 patients, stratified with relation to their level of asthma severity (25 patients for each level of severity - described by the GINA guidelines).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma confirmed by a pulmonologist
* Patient have had a lung function testing on the same day than the questionnaires are fulfilled.
* Age equal or upper than 18 years
* Agreement to participate to this study

Exclusion Criteria:

* Age under 18 years
* Refusal to participate to this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the consultation of pulmonology of a tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Level of asthma control | 1 day
  The five questionnaires are completed succesively on the same time.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU St Pierre; pulmonology department, Brussels, Belgium

REFERENCES:
- [Derived] Vermeulen F, de Meulder I, Paesmans M, Muylle I, Bruyneel M, Ninane V. Asthma control measurement using five different questionnaires: a prospective study. Respir Med. 2013 Sep;107(9):1314-21. doi: 10.1016/j.rmed.2013.07.003. Epub 2013 Jul 26. PMID 23890766